CLINICAL TRIAL: NCT00219219
Title: Zoledronic Acid in the Prevention of Skeletal-related Events in Hormone Refractory and Hormone-sensitive Prostate Cancer Patients With Bone Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Società Italiana di Urologia (SIU) (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EIT04
Record Dates: First submitted 2005-09-07; First posted 2005-09-22 (Estimated); Last update posted 2015-04-14 (Estimated); Status verified 2015-04

CONDITIONS: Prostate Cancer
Keywords: zoledronic acid; prostate cancer; SRE
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
The present study will give information about the course over time in skeletal-related events (SRE) in prostate cancer patients with bone metastases treated with zoledronic acid 4 mg administered as a 15-minute infusion every 4 weeks for a maximum of 15 infusions. The protocol will enroll patients with recent diagnosis of bone metastases from prostate cancer who are hormone-refractory, hormone-naïve or still hormone-sensitive, that represent the entire population of prostate cancer patients

ELIGIBILITY:
Inclusion Criteria

* Patients aged ≥18 years
* Written informed consent
* Histologically-proven prostate carcinoma
* ECOG performance status ≤ 2
* Life expectancy > 6 months
* Newly diagnosed (≤ 6 months prior to visit 1) bone metastases evidenced by bone scan or radiograph.
* Patients on androgen deprivation therapy (medical therapy with LHRH analogues + antiandrogens or surgical castration) or going to start it
* Patients with partners of childbearing potential should use a barrier method of contraception throughout the study

Exclusion Criteria

* Patients without a history of metastatic disease to the bone
* Prior treatment with bisphosphonates
* SREs prior to visit 2
* Prior treatment with calcitonin, mithramycin, or gallium nitrate within 2 weeks prior to baseline
* Corrected (adjusted for serum albumin - see Appendix 5 for the calculation) serum calcium concentration < 8.0 mg/dl (2.00 mmol/l)
* Serum creatinine concentration > 265 micromol/l (3.0 mg/dl) or a calculated creatinine clearance < 30 ml/minute or serious underlying renal disease or prior renal transplantation
* History of other malignant neoplasm within previous five years with exception of non-melanomatous skin cancer which has been satisfactorily treated
* Other known concurrent, severe medical disorder jeopardizing the life of the patient in the immediate future
* Patients treated with systemic investigational drug(s) and/or device(s) within the past 30 days or topical investigational drugs within the past 7 days
* Known hypersensitivity to zoledronic acid or other bisphosphonates
* History of noncompliance to medical regimens and patients who are considered potentially unreliable (for example drug or alchohol abusers) or incapable of giving informed consent as judged by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-09; Study Completion 2006-10

PRIMARY OUTCOMES:
occurence of skeletale related events (SREs) over time (time to first SRE,skeletal morbidity rate and proportion of patients experiencing SRE)

SECONDARY OUTCOMES:
Bone pain
Use of analgesic medication and ECOG performance status every three months
Bone specific alkaline phosphatase, serum N-telopeptide and parathyroid hormone will be evaluated after one month of treatment and then every three months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Bologna, Bologna, Italy